CLINICAL TRIAL: NCT03606252
Title: Specialized Proresolving Mediators Evaluation in Pneumocystis Pneumonia Human Infection : Pilot Study.
Brief Title: Specialized Proresolving Mediators in Pneumocystis Jirovecii Pneumonia
Acronym: INFLA-PCP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: RC31/18/0098; 2018-A01062-53 (Other: ID RCB)
Record Dates: First submitted 2018-07-19; First posted 2018-07-30 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Pneumonia, Pneumocystis
Keywords: Pneumocystis jirovecii; Pneumonia; Specialized Proresolving Mediators; Inflammation; prognosis
MeSH Terms: conditions — Pneumonia, Pneumocystis; Pneumonia; Inflammation | interventions — Blood Specimen Collection

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- pneumocystosis with favourable evolution (Other): patients with a favourable pneumocystosis outcome
  Interventions: Other: Blood sampling; Other: urine sampling
- pneumocystosis with unfavourable outcome (Other): patients with unfavourable pneumocystosis outcome
  Interventions: Other: Blood sampling; Other: urine sampling
- Pneumocystis colonization (Other): subject colonized by Pneumocystis jirovecii
  Interventions: Other: Blood sampling; Other: urine sampling

INTERVENTIONS:
Other: Blood sampling — 6 blood sample, 3 at J0 and 3 at J7 ( 2 tubes EDTA of 7mL, 1 tube Blood RNA of 3 mL)
Other: urine sampling — 2 urine sample (1 at J0 and 1 at J7)

SUMMARY:
This study aims to evaluate specialized proresolving mediators (SPM) concentrations for the first time in subjects infected with Pneumocystis jirovecii. SPM will be measured in blood and urine in patients with favourable or unfavourable outcome of Pneumocystis pneumonia and in patients colonized by Pneumocystis jirovecii. The hypothesis is that low levels of SPM in the blood could be predictive of a negative outcome of pneumocystosis.

DETAILED DESCRIPTION:
Pneumocystis pneumonia is a severe fungal disease threatening immunosuppressed subjects such as patients suffering from AIDS, oncohematological diseases or solid organ transplanted patients. The disease is characterized by an important inflammation in the infected lungs which is mainly responsible for lungs lesions. Despite an adequate treatment introduction, mortality is still around 20% which can not be explained by a treatment resistance. Specialized proresolving mediators (SPM), including lipoxins, maresins, protectins and resolvins, are newly described molecules implicated in the active process of inflammation resolution. The investigators hypothesis in this study is that high levels of SPM could be predictive of a good resolution of the harmful inflammation, thus a good evolution of the disease, in adequate pneumocystosis therapy conditions. On the contrary, low levels of SPM could be predictive of an unfavourable outcome despite a treatment targeting Pneumocystis jirovecii

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years old
* Patient with a social security cover.
* Free and informed oral consent given.
* Pneumocystis infection or colonization diagnosed on BAL (Broncho-alveolar liquid) or sputum at Toulouse University hospital Mycology laboratory.
* Adequate Pneumocystis therapy for infected patients (cotrimoxazole).

Exclusion Criteria:

* individuals placed under juridical protection,
* individuals placed under guardianship, or supervision.
* Pregnancy or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-03-12 (Actual); Study Completion 2020-03-12 (Actual)

PRIMARY OUTCOMES:
14,15-DHET blood level at the inclusio | Day 0
  variation of 14,15-DHET blood level at inclusion between each group
14,15-DHET blood level | Day 7
  variation of 14,15-DHET blood level at day 7 between each group

SECONDARY OUTCOMES:
14,15-DHET urine level | Day 0 and Day 7
  variation of 14,15-DHET urine level at inclusion ad day 7 between each group
Specialized Pro-Resolving Mediators in blood | Day 0 and Day 7
  Specialized Pro-Resolving Mediators in blood at inclusion and day 7 between each group
Specialized Pro-Resolving Mediators in urine | Day 0 and Day 7
  Specialized Pro-Resolving Mediators in urine at inclusion and day 7each between group
Expression levels of the SPM enzymes | Day 0 and day 7
  Expression levels of the enzymes implicated in SPM synthesis and catabolism in blood at D0 and day 7
Inflammatory blood profile | Day 0 and day 7
  Inflammatory blood profile with composite criteria pro-inflammatory and anti-inflammatory cytokines levels measured by flow cytometry
Immune cells profile | Day 0 and day 7
  immune cell proportions in blood measured by flow cytometry

CONTACTS AND LOCATIONS:
Overall Officials: Antoine Berry, PHD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Institut Fédératif de Biologie (IFB), CHU - Hôpital Purpan, Toulouse, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ko Y, Jeong BH, Park HY, Koh WJ, Suh GY, Chung MP, Kwon OJ, Jeon K. Outcomes of Pneumocystis pneumonia with respiratory failure in HIV-negative patients. J Crit Care. 2014 Jun;29(3):356-61. doi: 10.1016/j.jcrc.2013.12.005. Epub 2013 Dec 21. PMID 24440053
- [Background] Le Gal S, Robert-Gangneux F, Perrot M, Rouille A, Virmaux M, Damiani C, Totet A, Gangneux JP, Nevez G. Absence of Pneumocystis dihydropteroate synthase mutants in Brittany, France. Diagn Microbiol Infect Dis. 2013 May;76(1):113-5. doi: 10.1016/j.diagmicrobio.2013.01.018. Epub 2013 Feb 20. PMID 23433532
- [Background] Le Faouder P, Baillif V, Spreadbury I, Motta JP, Rousset P, Chene G, Guigne C, Terce F, Vanner S, Vergnolle N, Bertrand-Michel J, Dubourdeau M, Cenac N. LC-MS/MS method for rapid and concomitant quantification of pro-inflammatory and pro-resolving polyunsaturated fatty acid metabolites. J Chromatogr B Analyt Technol Biomed Life Sci. 2013 Aug 1;932:123-33. doi: 10.1016/j.jchromb.2013.06.014. Epub 2013 Jun 15. PMID 23831705
- [Background] Gilroy DW, Edin ML, De Maeyer RP, Bystrom J, Newson J, Lih FB, Stables M, Zeldin DC, Bishop-Bailey D. CYP450-derived oxylipins mediate inflammatory resolution. Proc Natl Acad Sci U S A. 2016 Jun 7;113(23):E3240-9. doi: 10.1073/pnas.1521453113. Epub 2016 May 25. PMID 27226306
- [Background] El Fane M, Sodqi M, Oulad Lahsen A, Chakib A, Marih L, Marhoum El Filali K. [Pneumocystosis during HIV infection]. Rev Pneumol Clin. 2016 Aug;72(4):248-54. doi: 10.1016/j.pneumo.2016.04.004. Epub 2016 Jun 24. French. PMID 27349824
- [Background] Colas RA, Shinohara M, Dalli J, Chiang N, Serhan CN. Identification and signature profiles for pro-resolving and inflammatory lipid mediators in human tissue. Am J Physiol Cell Physiol. 2014 Jul 1;307(1):C39-54. doi: 10.1152/ajpcell.00024.2014. Epub 2014 Apr 2. PMID 24696140
- [Background] Karsten E, Breen E, Herbert BR. Red blood cells are dynamic reservoirs of cytokines. Sci Rep. 2018 Feb 15;8(1):3101. doi: 10.1038/s41598-018-21387-w. PMID 29449599
- [Background] Keegan A, Charest K, Schmidt R, Briggs D, Deangelo DJ, Li B, Morgan EA, Pozdnyakova O. Flow cytometric minimal residual disease assessment of peripheral blood in acute lymphoblastic leukaemia patients has potential for early detection of relapsed extramedullary disease. J Clin Pathol. 2018 Jul;71(7):653-658. doi: 10.1136/jclinpath-2017-204828. Epub 2018 Mar 27. PMID 29588374